CLINICAL TRIAL: NCT01145391
Title: Health Promotion Outreach To Overcome Clinical Inertia In The Treatment Of Patients With Poorly-Controlled Hypertension
Brief Title: Reducing Clinical Inertia in Hypertension Treatment: A Pragmatic Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 09-0646
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; primary care; patient centered medical home; health information technology; clinical inertia
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients receive usual care.
- Intervention (Active Comparator): An outreach coordinator raised patient and provider awareness of unmet Blood Pressure goals, arranged Blood Pressure-focused clinic visits, and furnished providers with treatment decision support.
  Interventions: Other: Active Outreach to Patients and Providers

INTERVENTIONS:
Other: Active Outreach to Patients and Providers — An outreach coordinator raised patient and provider awareness of unmet Blood Pressure goals, arranged Blood Pressure-focused clinic visits, and furnished providers with treatment decision support.
  Arms: Intervention

SUMMARY:
The goal of this project is to use health information technology and team-based care in novel ways to support the establishment of a Patient-Centered Medical Home model of care aimed at improving the diagnosis and management of hypertension. Compared with patients who receive usual care, patients who receive intervention will have a lower average systolic blood pressure 9 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women age 18-79
* At least 2 Blood Pressure readings from separate days on record
* Average of last 3 Blood Pressure readings (or last 2 if only 2 available) with (Systolic Blood Pressure ≥140 or Diastolic Blood Pressure ≥90) and (last Systolic Blood Pressure ≥135 or last Diastolic Blood Pressure ≥85), recorded by any University of Colorado Hospital clinic within the last 18 months
* No clinic visit in the past month
* At least one Primary Care Physician visit in the past 18 months
* First Primary Care Physician visit at least 6 months in the past

Exclusion Criteria:

* Serious comorbidities, including active cancer diagnosis, hospice care, nursing home residence
* Diagnosis of diabetes (these patients are enrolled in a separate study that also targets Blood Pressure control)
* End-stage renal disease / hemodialysis
* Primary Care Physician appointment pending
* Patient instructed to monitor Blood Pressure at home / documentation of white coat hypertension
* Blood Pressure managed by specialist or outside provider

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Huebschmann, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Result] Huebschmann AG, Mizrahi T, Soenksen A, Beaty BL, Denberg TD. Reducing clinical inertia in hypertension treatment: a pragmatic randomized controlled trial. J Clin Hypertens (Greenwich). 2012 May;14(5):322-9. doi: 10.1111/j.1751-7176.2012.00607.x. Epub 2012 Mar 16. PMID 22533659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: September 2009 - January 2010. Types of locations: University of Colorado Hospital primary care clinics
Pre-assignment Details: Patients were excluded if they had serious comorbidities (e.g. active cancer diagnosis, hospice care, end-stage renal disease), diabetes mellitus, BP management by a nephrologist or other sub-specialist, a notation of white coat hypertension, or a notation that patient should monitor BP at home.
Groups:
- Intervention: An outreach coordinator raised patient and provider awareness of unmet BP goals, arranged BP-focused clinic visits, and furnished providers with treatment decision support.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 293 | 298
9 Months Post-randomization | 293 | 298
Completed | 293 | 298
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 293 | 298 | 591
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age, <45 years | 34.6 (6.4) | 35.5 (5.3) | 35.1 (5.8)
  Age, 45-54 years | 49.7 (2.8) | 49.9 (2.9) | 49.8 (2.8)
  Age, 55-64 years | 58.9 (3.0) | 59.6 (2.6) | 59.2 (2.8)
  Age, 65-79 years | 69.8 (3.9) | 69.6 (3.7) | 69.7 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 170 | 323
  Male | 140 | 128 | 268
Region of Enrollment [Number; unit: participants]
  United States | 293 | 298 | 591

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Hypothesis: compared with patients who receive usual care, patients who receive intervention will have an average systolic blood pressure that is at least 5 points lower 9 months after randomization.
Time Frame: Baseline, 9 months
Population: Intention-to-treat analyses using restricted maximum likelihood (REML) for a repeated measures model with incomplete data (SAS Proc Mixed). As this assumes that the occurrence of missing follow-up data depends only on observed data (i.e., pre-randomization values), we also performed a sensitivity analysis using the method proposed by Little.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Usual Care: Usual care
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 298 | 293
mm Hg | -10.1 (NA) [-12.2 to -8.0] | -9.1 (NA) [-11.3 to -6.8]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Non-Inferiority or Equivalence — Equivalence; p = 0.50, Mixed Models Analysis — For systolic blood pressure

2. Secondary Outcome: Clinical Inertia
Description: Definition of clinical inertia: failure of a primary care physician to initiate/intensify anti-hypertensive medications AND the failure to provide behavioral counseling to lower blood pressure during a clinic visit where blood pressure is elevated above 140/90 mm Hg. The clinical inertia measure is the percentage of clinic visits with clinical inertia present divided by the total number of clinic visits.
  We report a change in group mean levels of clinical inertia from baseline to 9 months post-randomization. Negative values for clinical inertia represent a decrease in the percentage of clinic visits where clinical inertia was present. Pre-randomization clinical inertia was assessed in the last 2 clinic visits prior to randomization, and post-randomization inertia was assessed in the first 2 post-randomization visits.
  Hypothesis: clinical inertia will be significantly greater in the usual care compared with intervention group in the post-randomization period.
Time Frame: Baseline, 9 months
Measure: Number (95% Confidence Interval); unit: % visits with inertia present
Arm/Group | Control | Intervention
Number analyzed (Participants) | 298 | 293
% visits with inertia present | -10.7 [-18.8 to -2.6] | -29.3 [-36.9 to -21.6]

ADVERSE EVENTS:
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 0/293 | 0/298
Other Adverse Events (participants affected / at risk) | 0/293 | 0/298

LIMITATIONS AND CAVEATS:
Adherence measures were not included. Patients with and without a formal diagnosis of hypertension were enrolled, but might require different intervention strategies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study funder, Novartis Pharmaceuticals Corporation, had no role in the data analysis or manuscript preparation; however, as part of the study agreement Novartis approved the investigators' study design and final manuscript.